CLINICAL TRIAL: NCT06211075
Title: Lay-guided Remotely Delivered Motivational Interviewing and Cognitive-behavioural Therapy for Insomnia: Protocol for a Feasibility and Pilot Study
Brief Title: Cracking the Code to Better Sleep: A Pioneering Study on Remote Support for Insomnia Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Overcome (Other)
Responsible Party: Principal Investigator, Tatiana Ermolenko, Lead Clinical Researcher, Overcome
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: P-PF-12.23.0001
Record Dates: First submitted 2023-11-29; First posted 2024-01-18 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Insomnia
Keywords: CBT-I; Motivational Interviewing; Insomnia; CBT for Insomnia; Mild Insomnia; Moderate Insomnia; CBT for Mild Insomnia; CBT for Moderate Insomnia; CBT for Mild/Moderate Insomnia; CBT-I for Mild Insomnia; CBT-I for Insomnia; CBT-I for Moderate Insomnia; Motivational Interviewing for Moderate Insomnia; Motivational Interviewing for Mild Insomnia; Motivational Interviewing for Insomnia; Feasibility of CBT-I; CBT-I pilot
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Group A (Experimental group, Intervention Group): will receive the intervention straight away Group B: (Control, Wait List Control Group): participants are allocated to the waitlist and will receive the intervention after the end of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The intervention will be delivered remotely via zoom or google meets, guided by Overcome coaches. Coaches are trained over two days via training slides, role plays and feedback. The intervention includes CBT-I and Motivational Interviewing.
  Interventions: Behavioral: Cognitive Behavioural Therapy for Insomnia with Motivational Interviewing
- Waitlist Control Group (WLC/WLCG) (No Intervention): Participants will receive the same benefits from the intervention after the end of the main study or after the last participant in the experimental group is interviewed at the post-intervention interview.

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy for Insomnia with Motivational Interviewing — This intervention implements elements of Cognitive Behavioural Therapy for Insomnia with motivational interview techniques incorporated into the intervention, aiming to build long-lasting motivation, better rapport with the patients and self-efficacy to increase engagement rate despite its remotely delivered format. The whole intervention is delivered online.
  Arms: Intervention Group

SUMMARY:
The goals of this clinical trial are to assess the feasibility of an internet-based Cognitive Behavioral Therapy for Insomnia (CBT-I) and Motivation Interviewing (MI) intervention for individuals aged 18 to 64 with mild to moderate insomnia, and/or mild anxiety/depression. The main questions it aims to answer are:

* Can internet-based CBT-I effectively improve sleep quality and reduce insomnia symptoms?
* Can internet-based CBT-I effectively improve sleep efficiency, sleep onset latency (SOL), and wake after sleep onset (WASO)?
* Is CBT-I treatment feasible to carry out remotely? What are the percentages of participants who dropped out of the study?
* Is internet-based CBT-I financially feasible compared to the traditional CBT-I intervention?

Eligible participants would be invited to participate in the research and randomised into two groups: Intervention and Waitlist Control. Both groups will have their baseline Insomnia Severity Index and Sleep Condition Indicator assessed prior to the main part of the research.

Participants in the Intervention group will go through 4 CBT-I sessions over the course of 4 weeks. These sessions will be delivered online by trained lay-person coaches, supervised directly by an experienced coach specialising in CBT-I. The Intervention group will also keep a sleep diary. At the end of the intervention, the investigators will interview 10 individuals to learn more about their experiences during the study.

Participants in the Waitlist Control Group will receive the same intervention after the end of the study. This group acts as a control for the Intervention group.

DETAILED DESCRIPTION:
The study discusses the prevalence and impact of insomnia, a sleep disorder affecting a significant portion of the population. Insomnia is linked to various health issues, including hypertension, obesity, depression, and reduced quality of life. Cognitive Behavioral Therapy for Insomnia (CBT-I) is recommended as an effective intervention, targeting maladaptive thoughts and behaviors related to sleep. Traditional CBT-I is delivered in a structured manner by licensed clinicians, but there are limitations to its accessibility and long-term efficacy. Internet-based CBT-I is proposed as a more accessible and convenient alternative, potentially overcoming the obstacles associated with traditional delivery methods. The intervention described in the text adopts a digital format, delivering CBT-I remotely with the inclusion of motivational interview techniques to enhance engagement and self-efficacy. Motivational Interviewing (MI) techniques aim to build motivation, rapport, and treatment adherence. MI has been successfully integrated into various treatment interventions, including addiction, psychotherapy, and suicide counselling. The text highlights the research gap in exploring the efficacy and feasibility of internet-based CBT-I, particularly for individuals with mild to moderate insomnia without comorbid disorders. Additionally, there is a lack of research on lay counselling in internet-based CBT-I. Investigating these areas can expand the accessibility and effectiveness of internet-based CBT-I for individuals suffering from insomnia.

This study aims to evaluate the effectiveness and feasibility of remotely delivered cognitive-behavioral therapy for insomnia (CBT-I) combined with motivational interviewing for individuals with mild-moderate insomnia. The efficacy of the treatment will be measured by changes in sleep efficiency, sleep onset latency (SOL), and wake after sleep onset (WASO) using sleep diaries, as well as improvements in sleep quality and insomnia symptoms measured by the Insomnia Severity Index (ISI) and Sleep Condition Indicator (SCI). The feasibility aspect of the study will explore participants' experiences and perceptions before and after the treatment, determine dropout rates and reasons for dropouts, and examine the frequency of incomplete sleep diary entries and the underlying reasons. The research questions to be answered include whether internet-based CBT-I can effectively improve sleep quality and reduce insomnia symptoms, improve sleep efficiency, SOL, and WASO, and whether remote CBT-I is feasible in terms of participant dropout rates and financial feasibility compared to traditional CBT-I interventions.

The British Association of Psychopharmacology (BAP) has updated guidelines for the treatment of insomnia in different settings, focusing on insomnia without comorbidity, or with mild depressive or anxiety symptoms. This paper aims to provide support for mild-moderate insomnia disorders. Comorbid insomnia and chronic insomnia disorders are better treated with a combination of cognitive behavioral therapy for insomnia (CBT-I) and pharmacological treatments. The inclusion criteria for the study include adults aged 18-64 with mild or no depression and mild anxiety symptoms, as measured by the PHQ-9 and GAD-7 questionnaires. Participants should also have self-reported difficulties initiating or maintaining sleep that align with the DSM-5 insomnia criteria. Exclusion criteria include severe or chronic insomnia, major psychiatric or neurological disorders, cognitive impairments, and current use of CBT-I or medication for insomnia. The initial screening process involves online self-report questionnaires (PHQ-9 & GAD-7) to identify potential participants. The PHQ-9 is used to assess depression symptoms, while the GAD-7 is used to screen for anxiety disorders. A score of 10 or higher on the PHQ-9 indicates probable depression, and a score of 8 or higher on the GAD-7 indicates probable anxiety disorder. The study will be conducted online, and participants will be recruited through the non-profit organization Overcome in the United Kingdom. Recruitment will involve advertisements on the Overcome website and social media, and interested individuals will complete the initial screening questionnaires via email. Eligible participants will be allocated either to the Intervention Group or Waitlist Control Group. The Intervention Group will receive information about their CBT-I coach and access to a sleep diary.

The study will focus on individuals with mild to moderate insomnia symptoms, as measured by the Insomnia Severity Index (ISI) score. Participants should not exhibit significant signs of clinical depression or anxiety. The CBT-I intervention will be delivered remotely via video conferencing, guided by trained coaches. The study will be conducted online, including participant recruitment, screening, informed consent, assessments, and group allocation. Outcome measures will be assessed online at baseline and one week after the intervention. A subset of participants will be invited to participate in qualitative process evaluation interviews. Participants will be recruited through an online registration process, and randomisation will be conducted to ensure a balanced distribution. The intervention will be delivered by a team of trained coaches, supervised by an experienced coach specialising in CBT-I. Data collection will occur at baseline and post-intervention.

The text discusses the analysis plan for a pilot study, focusing on descriptive analysis rather than hypothesis testing due to the absence of formal power calculations. The goal is to provide a detailed account of the collected data. The plan includes assessing data saturation, member checking, and triangulation to enhance the qualitative findings. The research team will maintain comprehensive records of screening, enrollment, completion of measures, and participation in sessions. Feasibility outcomes will be analysed using frequencies, proportions, means, and standard deviations. Feedback will be thematically analysed through audio-recorded interviews. For efficacy analysis, data will be exported to a software, where statistical analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-64
* PHQ-9 score 0-12 indicates no depression, mild or moderate depression
* GAD-7 score 0-12 indicates no anxiety, mild or moderate anxiety symptoms
* Individuals with self-reported difficulties initiating or maintaining sleep which are aligned with the DSM-5 insomnia criteria.
* Access to a computer or mobile with internet connectivity
* Ability to understand and speak English.
* Willingness and ability to participate in the internet-based CBT-I programme for five weeks (including the study-related assessments and post-follow-up interview)
* Willing to provide informed consent.

Exclusion Criteria:

* Individuals with a history of severe or chronic insomnia
* Those with a history of major psychiatric or neurological disorders (dementia, Alzheimer's disease)
* Those with cognitive impairments
* Those currently receiving or received CBT-I within the past year
* Those currently receiving medication for insomnia
* Individuals with known sleep disorders other than mild-moderate insomnia (sleep apnoea).
* Individuals suffering from chronic pain
* Pregnant and breastfeeding women.
* Not able to understand and respond in the study language.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-24 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Enrollment rate | From the beginning of recruitment until the first week of intervention.
  Number of people enrolled out of the number of people contacted. The higher percentage is the desirable outcome.
Eligibility rate | From the beginning of recruitment until the first week of intervention.
  Number of people eligible out of the number of people enrolled. The higher percentage is the desired outcome.
Attrition | From enrolment to post-intervention interview (5 weeks in total)
  Number of individuals who dropped out (dropouts only). The study aims to achieve lower attrition rates.
Change in Insomnia Severity Index (ISI) | From enrolment to post-intervention interview (5 weeks in total)
  The Insomnia Severity Index has seven questions. The seven answers are added up to get a total score. Total score categories are: 0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe). The questionnaire demonstrates positive test-retest reliability, internal consistency, and validity. Additionally, it is offered in three versions tailored for different perspectives: patient, clinician, and significant others (spouse). (Bastien et al., 2001; Morin et al., 2011)The lower scores signify milder insomnia. The study aims to achieve lowering in scores (baseline to post-intervention)
Change in Sleep Condition Indicator (SCI) | From enrolment to post-intervention interview (5 weeks in total)
  The questionnaire employs an eight-item rating scale, generating a severity score ranging from 0 to 32, where a higher score corresponds to better sleep. A score of 16 or lower suggests probable insomnia. Notably, the questionnaire demonstrates commendable internal consistency and concurrent validity, as evidenced by correlations with the PSQI and ISI. Its effectiveness extends to the measurement of daytime functioning. Furthermore, the questionnaire is accessible in various languages, attesting to its robust linguistic validation (Espie, et al., 2014; Wong et al, 2017). The lower scores signify milder insomnia. The study aims to achieve lowering in scores (baseline to post-intervention)
Adherence | From enrolment to post-intervention interview (5 weeks in total)
  Number of sleep diary entries and CBT-I sessions attended. The higher number is the desired outcome.

SECONDARY OUTCOMES:
Change in waketime self-reported by participants in their sleep diaries. | From enrolment to post-intervention interview (5 weeks in total)
  Participants will record their waketime every day for four weeks in their sleep diaries. The researchers will analyse the progression of the waketime over 4 weeks.
Change in Sleep Onset Latency (SOL) self-reported by participants in their sleep diaries. | From enrolment to post-intervention interview (5 weeks in total)
  Participants will record the duration of time from turning the light off to falling asleep in their sleep diaries over the course of intervention. The researchers will analyse the progression of SOL over 4 weeks. The lower the SOL, the better the outcomes are.
Change in Wake After Sleep Onset (WASO) self-reported by participants in their sleep diaries. | From enrolment to post-intervention interview (5 weeks in total)
  Participants will record their total number of minutes that a person is awake after having initially fallen asleep in their sleep diaries over the course of 4 weeks. The researchers will analyse the progression of SOL over 4 weeks. The lower the WASO, the better the outcomes are.
Change in 'perceived sleep quality' self-reported by participants in their sleep diaries. | From enrolment to post-intervention interview (5 weeks in total)
  Participants will report their perceived sleep quality every day in their sleep diaries. The will rate their sleep on the scale from 1 to 10. The researchers will analyse the progression of the scores over the course of 4 weeks and compare the scares from baseline assessment and post-intervention. The positive difference is the desired outcome.
Change in bedtime self-reported by participants in their sleep diaries | From enrolment to post-intervention interview (5 weeks in total)
  Participants will record their bedtime every day for four weeks in their sleep diaries. The researchers will analyse the progression of the bedtime over 4 weeks.
Change in number of naps from baseline to post-intervention. | From enrolment to post-intervention interview (5 weeks in total)
  Participants will record their number of naps every day for four weeks in their sleep diaries. The intervention aims to reduce the number of naps taken during the day over the course of the intervention.

OTHER OUTCOMES:
Satisfaction with the intervention | Post-intervention (Week 5)
  Participants will rate their satisfaction with the remotely delivered intervention (5-point Likert scale). The higher rates (7-10) are most desirable outcomes.
Perceived progress | Post-intervention (Week 5)
  Participants will rate the perceived progress in insomnia symptom management (10-point Likert scale). The higher rates (7-10) are most desirable outcomes.
Perceived adherence to the intervention | Post-intervention (Week 5)
  Participants will report their perceived adherence to the intervention (10-point Likert scale). The higher rates are the most desirable outcomes (7-10).

CONTACTS AND LOCATIONS:
Locations (1):
- Overcome, Arnside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
As it is a pilot and feasibility study, the researchers decided to not make the IPDs shareable to other researchers outside of Outcome. The access to trial IPD will be limited to the researchers within Overcome for future full-scale research. However, the researchers might reconsider at the end of the study, if the results from the thematic analysis and/or statistical analysis would be outside of our predictions.

REFERENCES:
- [Background] Yasugaki S, Okamura H, Kaneko A, Hayashi Y. Bidirectional relationship between sleep and depression. Neurosci Res. 2025 Feb;211:57-64. doi: 10.1016/j.neures.2023.04.006. Epub 2023 Apr 26. PMID 37116584
- [Background] Wilson SJ, Nutt DJ, Alford C, Argyropoulos SV, Baldwin DS, Bateson AN, Britton TC, Crowe C, Dijk DJ, Espie CA, Gringras P, Hajak G, Idzikowski C, Krystal AD, Nash JR, Selsick H, Sharpley AL, Wade AG. British Association for Psychopharmacology consensus statement on evidence-based treatment of insomnia, parasomnias and circadian rhythm disorders. J Psychopharmacol. 2010 Nov;24(11):1577-601. doi: 10.1177/0269881110379307. Epub 2010 Sep 2. PMID 20813762
- [Background] Theppornpitak W, Hemrungrojn S, Thienwiwatnukul K, Muntham D, Chirakalwasan N, Srisawart P. Effectiveness of internet-based CBT-I for the treatment of chronic subthreshold to moderate insomnia. Front Neurol. 2023 Jun 2;14:1180339. doi: 10.3389/fneur.2023.1180339. eCollection 2023. PMID 37346166
- [Background] Siengsukon CF, Alshehri M, Williams C, Drerup M, Lynch S. Feasibility and treatment effect of cognitive behavioral therapy for insomnia in individuals with multiple sclerosis: A pilot randomized controlled trial. Mult Scler Relat Disord. 2020 May;40:101958. doi: 10.1016/j.msard.2020.101958. Epub 2020 Jan 23. PMID 32014809
- [Background] Salwen-Deremer JK, Smith MT, Aschbrenner KA, Haskell HG, Speed BC, Siegel CA. A pilot feasibility trial of cognitive-behavioural therapy for insomnia in people with inflammatory bowel disease. BMJ Open Gastroenterol. 2021 Dec;8(1):e000805. doi: 10.1136/bmjgast-2021-000805. PMID 34969664
- [Background] Retzer L, Feil M, Reindl R, Richter K, Lehmann R, Stemmler M, Graessel E. Anonymous online cognitive behavioral therapy for sleep disorders in shift workers-a study protocol for a randomized controlled trial. Trials. 2021 Aug 16;22(1):539. doi: 10.1186/s13063-021-05437-9. PMID 34399824
- [Background] Pollak KI, Childers JW, Arnold RM. Applying motivational interviewing techniques to palliative care communication. J Palliat Med. 2011 May;14(5):587-92. doi: 10.1089/jpm.2010.0495. Epub 2011 Feb 3. PMID 21291329
- [Background] Plummer F, Manea L, Trepel D, McMillan D. Screening for anxiety disorders with the GAD-7 and GAD-2: a systematic review and diagnostic metaanalysis. Gen Hosp Psychiatry. 2016 Mar-Apr;39:24-31. doi: 10.1016/j.genhosppsych.2015.11.005. Epub 2015 Nov 18. PMID 26719105
- [Background] Matthews EE, Arnedt JT, McCarthy MS, Cuddihy LJ, Aloia MS. Adherence to cognitive behavioral therapy for insomnia: a systematic review. Sleep Med Rev. 2013 Dec;17(6):453-64. doi: 10.1016/j.smrv.2013.01.001. Epub 2013 Apr 17. PMID 23602124
- [Background] Karlin BE, Trockel M, Spira AP, Taylor CB, Manber R. National evaluation of the effectiveness of cognitive behavioral therapy for insomnia among older versus younger veterans. Int J Geriatr Psychiatry. 2015 Mar;30(3):308-15. doi: 10.1002/gps.4143. Epub 2014 May 29. PMID 24890708
- [Background] Johnson JA, Rash JA, Campbell TS, Savard J, Gehrman PR, Perlis M, Carlson LE, Garland SN. A systematic review and meta-analysis of randomized controlled trials of cognitive behavior therapy for insomnia (CBT-I) in cancer survivors. Sleep Med Rev. 2016 Jun;27:20-8. doi: 10.1016/j.smrv.2015.07.001. Epub 2015 Aug 1. PMID 26434673
- [Background] Grupp-Phelan J, Stevens J, Boyd S, Cohen DM, Ammerman RT, Liddy-Hicks S, Heck K, Marcus SC, Stone L, Campo JV, Bridge JA. Effect of a Motivational Interviewing-Based Intervention on Initiation of Mental Health Treatment and Mental Health After an Emergency Department Visit Among Suicidal Adolescents: A Randomized Clinical Trial. JAMA Netw Open. 2019 Dec 2;2(12):e1917941. doi: 10.1001/jamanetworkopen.2019.17941. PMID 31860104
- [Background] Glass J, Lanctot KL, Herrmann N, Sproule BA, Busto UE. Sedative hypnotics in older people with insomnia: meta-analysis of risks and benefits. BMJ. 2005 Nov 19;331(7526):1169. doi: 10.1136/bmj.38623.768588.47. Epub 2005 Nov 11. PMID 16284208
- [Background] Espie CA, Kyle SD, Williams C, Ong JC, Douglas NJ, Hames P, Brown JS. A randomized, placebo-controlled trial of online cognitive behavioral therapy for chronic insomnia disorder delivered via an automated media-rich web application. Sleep. 2012 Jun 1;35(6):769-81. doi: 10.5665/sleep.1872. PMID 22654196
- [Background] Edinger JD, Bonnet MH, Bootzin RR, Doghramji K, Dorsey CM, Espie CA, Jamieson AO, McCall WV, Morin CM, Stepanski EJ; American Academy of Sleep Medicine Work Group. Derivation of research diagnostic criteria for insomnia: report of an American Academy of Sleep Medicine Work Group. Sleep. 2004 Dec 15;27(8):1567-96. doi: 10.1093/sleep/27.8.1567. PMID 15683149
- [Background] Dunn C, Deroo L, Rivara FP. The use of brief interventions adapted from motivational interviewing across behavioral domains: a systematic review. Addiction. 2001 Dec;96(12):1725-42. doi: 10.1046/j.1360-0443.2001.961217253.x. PMID 11784466
- [Background] Costantini L, Pasquarella C, Odone A, Colucci ME, Costanza A, Serafini G, Aguglia A, Belvederi Murri M, Brakoulias V, Amore M, Ghaemi SN, Amerio A. Screening for depression in primary care with Patient Health Questionnaire-9 (PHQ-9): A systematic review. J Affect Disord. 2021 Jan 15;279:473-483. doi: 10.1016/j.jad.2020.09.131. Epub 2020 Oct 6. PMID 33126078
- [Background] Christensen DL, Braun KVN, Baio J, Bilder D, Charles J, Constantino JN, Daniels J, Durkin MS, Fitzgerald RT, Kurzius-Spencer M, Lee LC, Pettygrove S, Robinson C, Schulz E, Wells C, Wingate MS, Zahorodny W, Yeargin-Allsopp M. Prevalence and Characteristics of Autism Spectrum Disorder Among Children Aged 8 Years - Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2012. MMWR Surveill Summ. 2018 Nov 16;65(13):1-23. doi: 10.15585/mmwr.ss6513a1. PMID 30439868
- [Background] Cassel M, Blom K, Gatzacis J, Renblad P, Kaldo V, Jernelov S. Clinical feasibility of cognitive behavioural therapy for insomnia in a real-world mixed sample at a specialized psychiatric outpatient clinic. BMC Psychiatry. 2022 Sep 9;22(1):600. doi: 10.1186/s12888-022-04231-4. PMID 36085009
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Bertisch SM, Pollock BD, Mittleman MA, Buysse DJ, Bazzano LA, Gottlieb DJ, Redline S. Insomnia with objective short sleep duration and risk of incident cardiovascular disease and all-cause mortality: Sleep Heart Health Study. Sleep. 2018 Jun 1;41(6):zsy047. doi: 10.1093/sleep/zsy047. PMID 29522193
- [Background] undefined
- [Background] Alimoradi Z, Jafari E, Brostrom A, Ohayon MM, Lin CY, Griffiths MD, Blom K, Jernelov S, Kaldo V, Pakpour AH. Effects of cognitive behavioral therapy for insomnia (CBT-I) on quality of life: A systematic review and meta-analysis. Sleep Med Rev. 2022 Aug;64:101646. doi: 10.1016/j.smrv.2022.101646. Epub 2022 May 10. PMID 35653951